CLINICAL TRIAL: NCT00127803
Title: A Phase I Randomized, Placebo-Controlled, Double-Blind, Dose-Ranging Study of the Safety, Tolerability and Immunogenicity of a Clostridium Difficile Toxoid Vaccine, Alum Adsorbed, in Healthy Adult Volunteers (18-55 Years)
Brief Title: Safety, Tolerability, and Immunogenicity Study of a Clostridium Difficile Toxoid Vaccine in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: H-030-008
Record Dates: First submitted 2005-08-05; First posted 2005-08-09 (Estimated); Results first posted 2012-05-21 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-09

CONDITIONS: Clostridium Infections
Keywords: Clostridium difficile
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Participants will receive a dose of vaccine diluent (placebo) on Days 0, 28, and 56, respectively.
  Interventions: Biological: Placebo (vaccine diluent)
- Low dose vaccine (Experimental): Participants will receive a 2 μg dose of C. difficile toxoid vaccine on Days 0, 28, and 56, respectively.
  Interventions: Biological: Clostridium difficile vaccine
- Medium dose vaccine (Experimental): Participants will receive a 10 μg dose of C. difficile toxoid vaccine on Days 0, 28, and 56, respectively
  Interventions: Biological: Clostridium difficile vaccine
- High dose vaccine (Experimental): Participants will receive a 50 μg dose of C. difficile toxoid vaccine on Days 0, 28, and 56, respectively
  Interventions: Biological: Clostridium difficile vaccine

INTERVENTIONS:
Biological: Placebo (vaccine diluent) — 0.5 mL, intramuscular (IM) on Days 0, 28, and 56, respectively.
  Arms: Placebo
Biological: Clostridium difficile vaccine — 0.5 mL, intramuscular on Days 0, 28, and 56, respectively.
  Arms: Low dose vaccine
Biological: Clostridium difficile vaccine — 0.5 mL, intramuscular on Days 0, 28, and 56, respectively.
  Arms: Medium dose vaccine
Biological: Clostridium difficile vaccine — 0.5 mL, intramuscular on Days 0, 28, and 56, respectively.
  Arms: High dose vaccine

SUMMARY:
The purpose of this study is to determine the safety and tolerability of a modified C. difficile vaccine at 3 dose levels compared with a placebo control administered via intramuscular injection in healthy adults aged 18-55 years of age.

DETAILED DESCRIPTION:
Clostridium difficile is the leading infectious cause of nosocomial diarrhea in developed countries. Hospital outbreaks of Clostridium difficile-associated diarrhea (CDAD) are associated with substantial patient morbidity and mortality. Conventional therapy with antibiotics often results in secondary infection with resistant organisms or clinical relapse after discontinuation of the antimicrobial course. New strategies are needed to limit the impact of this opportunistic pathogen. Considerable evidence exists that immunity against C. difficile toxins may be effective in controlling CDAD. 48 subjects will be enrolled to receive one of three dose levels of modified C difficile vaccine or placebo administered on a 3-dose schedule. The study consists of a 30-day screening period, a 70-day treatment period, one follow-up phone interview 2 months after the last vaccination, and one follow-up clinic visit 6 months after the last vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Adult males or females, 18-55 years (inclusive)
* In good general health
* Clinical lab tests within normal range
* Non-pregnant female subjects
* Able and willing to participate for duration of study and must not participate in any other experimental study for at least 60 days after receiving the last dose of study vaccine

Exclusion Criteria:

* Evidence of C. difficile infection
* Evidence of any previous antibiotic-associated diarrhea
* Active or inactive inflammatory bowel disease, irritable colon syndrome, chronic abdominal pain or other chronic diarrhea
* History of malignancy within 5 years
* History of anaphylaxis, asthma or severe vaccine or severe allergic drug reaction
* Known or suspected history of immunodeficiency;
* Active or inactive immune-mediated or inflammatory disease;
* Pregnant or lactating female subjects;
* History of drug or alcohol abuse disorders;
* Serology positive for HIV, hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV)
* Receipt of antibiotic therapy or an investigational drug within prior 30 days
* Blood or organ donation within prior 30 days

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2005-07; Primary Completion 2006-01 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Marbury, MD, Principal Investigator — Orlando Clinical Research Center; Richard Greenberg, MD, Principal Investigator — University of Kentucky

REFERENCES:
- [Derived] Greenberg RN, Marbury TC, Foglia G, Warny M. Phase I dose finding studies of an adjuvanted Clostridium difficile toxoid vaccine. Vaccine. 2012 Mar 16;30(13):2245-9. doi: 10.1016/j.vaccine.2012.01.065. Epub 2012 Feb 2. PMID 22306375
- See also: Related Info — http://www.sanofipasteur.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 13 July 2005 to 27 July 2005 in 2 medical centers in the US.
Pre-assignment Details: A total of 50 participants who met the inclusion, but no exclusion criteria were enrolled and vaccinated.
Groups:
- Placebo Group: Participants who received 3 doses of vaccine diluent (placebo) on Days 0, 28, and 56.
- Low Dose Vaccine Group: Participants who received 3 doses of vaccine containing 2 μg C. difficile toxoid on Days 0, 28, and 56.
- Medium Dose Vaccine Group: Participants who received 3 doses of vaccine containing 10 μg C. difficile toxoid on Days 0, 28, and 56.
- High Dose Vaccine Group: Participants who received 3 doses of vaccine containing 50 μg C. difficile toxoid on Days 0, 28, and 56.
Period: Overall Study
Arm/Group | Placebo Group | Low Dose Vaccine Group | Medium Dose Vaccine Group | High Dose Vaccine Group
Started | 13 | 13 | 12 | 12
Completed | 10 | 13 | 12 | 11
Not Completed | 3 | 0 | 0 | 1
Not completed — Adverse Event | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Group | Low Dose Vaccine Group | Medium Dose Vaccine Group | High Dose Vaccine Group | Total
Number analyzed (Participants) | 13 | 13 | 12 | 12 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 12 | 12 | 50
  >=65 years | 0 | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: Years] | 33.6 (12.49) | 30.8 (10.26) | 30.4 (9.78) | 32.6 (9.07) | 31.9 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 6 | 8 | 9 | 33
  Male | 3 | 7 | 4 | 3 | 17
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 12 | 12 | 50

OUTCOME MEASURES:

1. Secondary Outcome: Number of Participants With Seroconversion for Toxin A and Toxin B Post-vaccination With Either One of Three Formulations of the Clostridium Difficile Vaccine or a Placebo Vaccine.
Description: Seroconversion was defined as a ≥4-fold increase in antibody levels from Baseline. For values below the limit of quantification (LLQ) for the assay, the LLQ was used.
  Serum anti-toxin IgG levels were determined by enzyme linked immunosorbent assay (ELISA).
Time Frame: Days 28, 56, 70, and 236 Post First Vaccination
Population: Serum anti-toxin levels were assessed in the Fully Evaluable (Per-Protocol) Population.
Measure: Number; unit: Participants
Arm/Group | Placebo Group | Low Dose Vaccine Group | Medium Dose Vaccine Group | High Dose Vaccine Group
Number analyzed (Participants) | 10 | 13 | 12 | 11
Participants
  Toxin A Day 28 | 0 | 6 | 5 | 10
  Toxin A Day 56 | 0 | 13 | 12 | 11
  Toxin A Day 70 | 0 | 13 | 12 | 11
  Toxin A Day 236 | 0 | 12 | 12 | 10
  Toxin B Day 28 | 0 | 2 | 5 | 7
  Toxin B Day 56 | 0 | 3 | 6 | 7
  Toxin B Day 70 | 0 | 6 | 7 | 8
  Toxin B Day 236 | 0 | 2 | 4 | 6

2. Primary Outcome: Number of Participants Reporting Solicited Injection Site Erythema and Tenderness Post-vaccination With Either One of Three Formulations of Clostridium Difficile Vaccines or a Placebo Vaccine.
Time Frame: Day 0 and up to 7 days post each vaccination
Population: Safety assessments were on the safety population.
Measure: Number; unit: Participants
Arm/Group | Placebo Group | Low Dose Vaccine Group | Medium Dose Vaccine Group | High Dose Vaccine Group
Number analyzed (Participants) | 13 | 13 | 12 | 12
Participants
  Erythema Day 0 | 2 | 0 | 1 | 2
  Erythema Day 28 | 0 | 3 | 3 | 2
  Erythema Day 56 | 2 | 2 | 3 | 3
  Tenderness Day 0 | 0 | 0 | 3 | 1
  Tenderness Day 28 | 0 | 1 | 0 | 2
  Tenderness Day 56 | 0 | 2 | 1 | 1

3. Primary Outcome: Number of Participants Reporting Treatment-Emergent Adverse Events Post-vaccination With Either One of Three Formulations of the Clostridium Difficile Vaccine or a Placebo Vaccine.
Time Frame: Day 0 to up to 70 days post-first vaccination
Population: Safety assessments were on the safety population.
Measure: Number; unit: Participants
Arm/Group | Placebo Group | Low Dose Vaccine Group | Medium Dose Vaccine Group | High Dose Vaccine Group
Number analyzed (Participants) | 13 | 13 | 12 | 12
Participants
  Injection site pain | 8 | 11 | 11 | 12
  Injection site erythema | 2 | 6 | 5 | 6
  Red blood cells urine positive | 2 | 5 | 6 | 5
  Protein urine present | 2 | 6 | 4 | 5
  Eosinophil count increased | 1 | 2 | 5 | 3
  Headache | 4 | 4 | 3 | 0
  Upper respiratory tract infection | 2 | 3 | 2 | 3
  White blood cells urine positive | 3 | 1 | 3 | 3
  Pain in extremity | 5 | 0 | 1 | 3
  Injection site swelling | 1 | 2 | 3 | 3
  Diarrhoea | 3 | 2 | 0 | 3
  Blood urea increased | 0 | 1 | 4 | 2
  Injection site induration | 0 | 1 | 4 | 2
  Abdominal pain | 1 | 0 | 1 | 4
  Injection site warmth | 1 | 1 | 1 | 3
  Fatigue | 2 | 1 | 1 | 2
  Myalgia | 2 | 1 | 1 | 1
  Injection site pruritus | 0 | 0 | 1 | 3
  White blood cell count decreased | 0 | 0 | 2 | 2
  Blood potassium increased | 3 | 1 | 0 | 0
  Sensation of heaviness | 0 | 0 | 1 | 2
  Injection site irritation | 2 | 0 | 1 | 0
  Sinus headache | 0 | 2 | 0 | 0
  White blood cell count increased | 0 | 2 | 0 | 0
  Blood potassium increased | 3 | 1 | 0 | 0
  Injection site paraesthesia | 2 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination for up to 1 year post-vaccination.
Arm/Group | Placebo Group | Low Dose Vaccine Group | Medium Dose Vaccine Group | High Dose Vaccine Group
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 13/13 | 13/13 | 12/12 | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Placebo Group (N=13) | Low Dose Vaccine Group (N=13) | Medium Dose Vaccine Group (N=12) | High Dose Vaccine Group (N=12)
Eyelid cyst (Eye disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 0 | 3
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Asthenia (General disorders) | 1 | 0 | 1 | 0
Fatigue (General disorders) | 2 | 1 | 1 | 2
Induration (General disorders) | 1 | 0 | 0 | 0
Injection site anaesthesia (General disorders) | 1 | 1 | 0 | 0
Injection site discomfort (General disorders) | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 2 | 6 | 5 | 6
Injection site haemorrhage (General disorders) | 1 | 0 | 1 | 1
Injection site induration (General disorders) | 0 | 1 | 4 | 2
Injection site irritation (General disorders) | 2 | 0 | 1 | 0
Injection site oedema (General disorders) | 0 | 0 | 0 | 1
Injection site pain (General disorders) | 8 | 11 | 11 | 12
Injection site paraesthesia (General disorders) | 2 | 0 | 0 | 0
Injection site pruritus (General disorders) | 0 | 0 | 1 | 3
Injection site swelling (General disorders) | 1 | 2 | 3 | 3
Injection site warmth (General disorders) | 1 | 1 | 1 | 3
Malaise (General disorders) | 1 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 3 | 2 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Blood bilirubin increased (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Blood calcium increased (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Blood creatinine increased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Blood potassium decreased (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1
Blood potassium increased (Blood and lymphatic system disorders) | 3 | 1 | 0 | 0
Blood urea increased (Blood and lymphatic system disorders) | 0 | 1 | 4 | 2
Eosinophil count increased (Blood and lymphatic system disorders) | 1 | 2 | 5 | 3
Lymphocyte count decreased (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Protein urine present (Blood and lymphatic system disorders) | 2 | 6 | 4 | 5
Red blood cell count increased (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Red blood cells urine positive (Blood and lymphatic system disorders) | 2 | 5 | 6 | 5
Transaminase increased (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
White blood cell count decreased (Blood and lymphatic system disorders) | 0 | 0 | 2 | 2
White blood cell count increased (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
White blood cells urine positive (Blood and lymphatic system disorders) | 3 | 1 | 3 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 0 | 1 | 3
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 2
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 4 | 3 | 0
Sinus headache (Nervous system disorders) | 0 | 2 | 0/0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0
Nervousness (Psychiatric disorders) | 1 | 0 | 0 | 0
Metorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1/2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications